CLINICAL TRIAL: NCT05346614
Title: Digital, Blended Lifestyle Intervention Program for Remission and Improved Management of Type 2 Diabetes
Brief Title: Digital, Blended Lifestyle Intervention for Type 2 Diabetes Remission
Acronym: IBIDEM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ancora Health B.V. (Industry)
Collaborators: University of Groningen (Other); Universiteit Leiden (Other); TNO (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL77688.056.21
Record Dates: First submitted 2022-02-03; First posted 2022-04-26 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This a randomized intervention study. Subjects will be randomly allocated using a 5:1 ratio between the control and intervention groups.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to the treatment allocations. It is not possible to blind participants or care providers who will be providing the intervention, as this is a lifestyle intervention. Controls receive usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active lifestyle intervention (Experimental): Individuals in the active intervention group will undergo diabetyping (diabetes type 2 phenotyping: glucose, and C-peptide responses to a glucose challenge). Based on the diabetype, individuals will receive recommendations to follow either a calorie-restricted (500kcal deficit minimum) low carbohydrate or a modified Mediterranean diet for a period of 18 weeks (total intervention is 24 weeks). Secondly, individuals will follow a personalized exercise program. Guidance and coaching (individual and small group) will be given via mobile app and digital platform. Individuals will receive real-time feedback based on their diet, exercise, and glucose levels (via continuous glucose monitoring for 4 weeks). Medications will be slowly withdrawn over the intervention period, with a focus on the first phase of the intervention.
  Interventions: Behavioral: Lifestyle intervention
- Usual care group (No Intervention): Individuals in the usual care group will receive standard diabetes care.

INTERVENTIONS:
Behavioral: Lifestyle intervention — Lifestyle coaching will be given on a digital app-based platform. Individuals will receive real-time feedback via a smart scale, activity monitor, and continuous glucose monitor (first 4 weeks, longer if required). Coaching will be focused on gradual behavior change, assisted by digital nudges, one-on-one, and small group coaching sessions. Coaching will include education regarding lifestyle to improve health literacy with respect to diet and diabetes management. Additionally, coaches will guide participants in the implementation of individualized diet and exercise program with varying levels of carbohydrate restriction and caloric deficit.
  Arms: Active lifestyle intervention

SUMMARY:
410 Dutch type 2 diabetes patients will be randomized using a 5:1 ratio to intervention group versus control, to a lifestyle intervention program given via a mobile application and digital platform. Active participants will undergo diabetyping, where blood glucose and c-peptide responses to a glucose challenge are measured, and be recommended to follow a calorie-restricted (minimum 500 kcal deficit) low-carbohydrate, or restricted carbohydrate (120g) Mediterranean diet and customized exercise program for a period of 24 weeks. Individuals will then be followed for a period of 2 years following the intervention.

DETAILED DESCRIPTION:
Patients will partake in a 24-week intervention followed by a two-year follow-up period. The intervention will consist of diabetic phenotyping (diabetyping), and a personalized app-based lifestyle intervention, done in conjunction with usual care, the so-called blended care model. Individuals will be allocated to either a high (unsaturated) fat, low-carbohydrate Mediterranean (50 g), or the Mediterranean with limited carbohydrates (120 g) diet based on their diabetype, insulin use, and personal preference. This will be given in conjunction with physical activity program, which will focus more on aerobic activity or resistance training depending on diabetype. All participants will be provided with additional coaching to support behavioral change, which will include aspects of diet, physical activity but also aspects of mindfulness, and emotion regulation. The participants will be assessed at screening, before the start of the maintenance phase, and at follow-ups one, two, and three. Control patients will follow the usual care and will also be followed up, following the same schedule. The treatment is further clarified below:

Prior to commencing the study, participants in the active intervention group will receive a kit containing all the necessary products (i.e. wearable, smart scale, and glucose monitor), information, and instructions (where applicable) for participating in the study. Moreover, they will be carefully informed about the types of personalisations available to them. The participants will have either a whole food type diet or a low carbohydrate diet recommended to them based on their metabolic profiles. In addition, they will also have specific types of exercise recommended to them. Participants' treating physicians and coaches will be informed about their choices, and will receive supporting medication adjustment documents, based on those made in previous studies. It will remain the responsibility of the treating physicians to adjust any medications the participants are receiving.

The control group is required to meet the same criteria as the intervention group. The control group only receives health assessments (with the exception of the diabetyping), and will not receive any health intervention. They will continue to receive standard diabetes care.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes: Diagnosis of T2DM without physician defined end-organ failure
* BMI: 25 to 45 kg/m²
* Age: 18 to 75 years
* Most recent HbA1c value should be greater than 6.0% (>43 mmol/mol); if less than 6.5% (<48 mmol/mol), individuals should still be receiving anti-diabetic medication
* Tech-savvy (patients are required to be able to fully use smartphone or tablet)
* Display interest and motivation to enroll in a digital, lifestyle intervention for diabetes

Exclusion Criteria:

* Weight loss of more than five kg or greater than 10% within the past six months
* Serious co-morbidities, for example, a severe form of chronic obstructive pulmonary disease (Gold III or IV), bariatric surgery, heart failure (classes 2-4) kidney failure, or another medically determined end-stage organ failure
* Substance abuse
* Learning difficulties limiting the participation in a digital health intervention and or limiting the comprehension of trial goals or coaching curriculum.
* Current treatment with anti-obesity drugs
* Pregnancy, consideration of pregnancy within the study period, lactation or having given birth within the previous nine months
* Hospital admission for depression
* Major psychiatric disorder (e.g., schizophrenia, bipolar disorder) or use of antipsychotic drugs.
* Currently uncontrolled or eating disorder or purging behavior
* Type 1 diabetes
* History of keto-acidosis
* Myocardial infarction, stroke, angina, or coronary insufficiency within the previous six months
* Diabetic retinopathy requiring treatment
* Creatinine > 2.0 mg·dL-1 or > 152.5 µmol·L-1
* Urinary albumin > 1 g·dL-1 or > 10 g·L-1
* Cancer requiring treatment in the past five years, with the exception of non-melanoma skin cancer
* Chronic infectious disease requiring ongoing treatment
* Other chronic diseases or conditions likely to limit lifespan to less than six years
* Severe visual impairment or other impairment preventing interaction with digital content
* Non-English or Non-Dutch speaking
* Excessive alcohol intake (acute or chronic) defined as the average consumption of three or more alcohol-containing beverages daily or consumption of more than 14 alcoholic beverages per week
* Cholelithiasis or biliary dysfunction
* Use of an insulin pump
* Participation in diabetes therapy within the preceding three years; participation in concurrent weight management or interventional research protocol,
* Untreated thyroid disease,
* Requirement of a prescribed medical diet
* A recent on-record estimated glomerular filtration rate of less than 30 mL/min per 1.732 m²
* Incapacitated patients, and thus unable to fully participate in the trial.
* uncontrolled blood pressure (SBP > 170 mmHg and/or DBP > 100 mmHg)
* For nutritional ketosis specifically: impaired hepatic function (Bilirubin >2 mg·dL-1 or >34.2 µmol·L-1, Albumin < 3.5 g·dL-1 or <35 g·L-1)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of diabetes remission | 1 year
  Percentage of patients achieving complete diabetes remission. Diabetes remission rates amongst the active intervention group will be reported as the number of participants who have achieved fasting glucose < 7 mmol/L or HbA1c < 6.5% (48 mmol/mol) on two separate occasions 6 months apart, and glucose-lowering therapy has been stopped.

SECONDARY OUTCOMES:
Rates of improved glycaemic control | Will be reported at all follow-up moments (6 months, 1 year, and 2 years)
  Percentage of patients achieving improved glycaemic control. This will be defined as the number of individuals who achieve a reduction in glycated hemoglobin (HbA1c), and or reduced dependence on glucose-lowering medications, defined as the number of medications or dose.
Blood lipids | Will be reported at all follow-up moments (6 months, 1 year, and 2 years)
  Changes in blood lipids, namely triglycerides, total cholesterol, LDL, and HDL will be measured as an indicator of health status
Weight loss | Will be reported at all follow-up moments (6 months, 1 year, and 2 years)
  Weight loss will be measured as change in weight compared to baseline. It will be measured as an indicator of participant compliance and feasibility of the program.
Remission versus diabetype | Will be reported at all follow-up moments (6 months, 1 year, and 2 years)
  The association between diabetype* as determined by response to an oral glucose tolerance test with remission will be determined
  * de Hoogh IM, Oosterman JE, Otten W, et al. The Effect of a Lifestyle Intervention on Type 2 Diabetes Pathophysiology and Remission: The Stevenshof Pilot Study. Nutrients 2021;13(7):2193.
Cost effectiveness | Will be reported at all follow-up moments (6 months, 1 year, and 2 years)
  The cost of the intervention will be analyzed in comparison with that of usual care, in terms of doctor and hospital visits, as well as the use of supportive medical care ex. physiotherapy.
Digital engagement as measured by the Engagement Index | Up to 1 year
  Digital engagement will be digitally recorded as an engagement index, which is based on the frequency of user engagement with the app and digital content.
Compliance | Up to 1 year
  Compliance will be assessed as a score based on the user's participation and success in coaching activities, educational sessions, and diet, physical activity and blood sugar measurement logging goals.

CONTACTS AND LOCATIONS:
Overall Officials: Suzan Wopereis, PhD, Principal Investigator — TNO; Maarten van Aken, MD PhD, Principal Investigator — Haga Ziekenhuis; Elly Vogelzang, MD, Principal Investigator — Center Medische Kwartier Eindhoven; Janet Kist, MD, Principal Investigator — Huisartsenpraktijk Zonneoord; Jan Hoogsteen, MD, Principal Investigator — Ancora Health; Rimke Vos, PhD, Principal Investigator — Department of Public Health and Primary Care / LUMC-Campus Den Haag
Locations (4):
- Netherlands (4):
  - St. Anna Ziekenhuis, Eindhoven, Limburg
  - Center Medische Kwartier Eindhoven, Eindhoven, North Brabant
  - Huisartsenpraktijk Zonneoord, The Hague, South Holland
  - Haga Ziekenhuis, The Hague, South Holland

IPD SHARING:
Plan to Share IPD: Yes
The data will be made available to researchers upon motivated request. Moreover, all supporting documents will be submitted upon publication of the study protocol and results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Undecided.
Access Criteria: Undecided.